CLINICAL TRIAL: NCT00975611
Title: Amantadine Addition to Paliperidone ER or Risperidone Consta Therapy for Prolactin Elevation
Brief Title: Study of Amantadine for Risperidone Consta or Paliperidone Treated Patients to Decrease Prolactin Elevation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The sponsor withdrew support due to slow accrual of eligible subjects.
Sponsor: David C. Henderson, MD (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor-Investigator, David C. Henderson, MD, Associate Professor, North Suffolk Mental Health Association
Organization: North Suffolk Mental Health Association (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R076477PD14002
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; paliperidone ER; risperidone Consta; prolactin; hyperprolactinemia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hyperprolactinemia | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Amantadine 100mg BID (Active Comparator): Subjects take amantadine 100mg tablets twice per day (BID)
  Interventions: Drug: Amantadine Hydrochloride, USP
- Amantadine, 200mg BID (Active Comparator): Subjects take amantadine 200mg tablets twice per day (BID)
  Interventions: Drug: Amantadine Hydrochloride, USP
- Amantadine, placebo BID (Placebo Comparator): Subjects take placebo tablets twice per day (BID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amantadine Hydrochloride, USP — amantadine tablets 100 mg. BID for 4 weeks
  Other Names: Symmetrel
  Arms: Amantadine 100mg BID
Drug: Amantadine Hydrochloride, USP — amantadine 200 mg. tablets BID for 4 weeks
  Other Names: Symmetrel
  Arms: Amantadine, 200mg BID
Drug: Placebo — tablets BID, for 4 weeks
  Other Names: Symmetrel placebo
  Arms: Amantadine, placebo BID

SUMMARY:
The purpose of this study is to show that amantadine might help to reduce the side effect of the medications which are prescribed to treat schizophrenia or schizoaffective disorder. High level of hormone prolactin, or hyperprolactinemia, is one of the side effects which might be developed in patients treated with the paliperidone ER or risperidone Consta.

High level of prolactin might stimulate breast development, might decrease sexual desire (libido). The goals of this study are to demonstrate that amantadine lowers prolactin levels, decreases side effects, and improves psychiatric symptoms.

DETAILED DESCRIPTION:
Trial Description: A double-blind, placebo-controlled, prospective, randomized trial to evaluate the effects of two doses of amantadine or placebo in the management of antipsychotic-induced hyperprolactinemia and psychiatric status in patients with schizophrenia or schizoaffective disorder who are clinically stable on paliperidone ER or risperidone Consta. Placebo or amantadine 100 mg or 200 mg BID will be administered to participants for 4 consecutive weeks as an adjunctive therapy in 72 schizophrenia subjects treated with paliperidone or risperidone Consta to examine amantadine effects on fasting AM serum prolactin levels. Participants will be followed after suspension of amantadine or placebo for an additional 4 weeks for safety purposes. The goals of this study are to prospectively demonstrate that amantadine lowers prolactin levels, and evaluate the impact of amantadine on psychiatric symptoms, and on prolactin-related side effects in patients treated with paliperidone ER or risperidone Consta.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-65 years
* Diagnosis of schizophrenia, schizoaffective disorder, any subtype or schizophreniform disorder
* Well established compliance with out-patient medications including paliperidone ER or risperidone Consta for 3 months

Exclusion Criteria:

* Current substance or alcohol abuse
* Significant medical illness
* Women who are pregnant, breastfeeding, or who are unwilling or unable to use an effective form of birth control during the entire study
* Subjects treated with more than one antipsychotic drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C. Henderson, M.D., Principal Investigator — North Sufflok Mental Health Association, Freedom Trail Clinic
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Freedom Trail Clinic, MGH Schizophrenia Program
Pre-assignment Details: Of the 22 consented subjects, 15 screen-failed because prolactin levels did not meet eligibility criteria, and 1 screen failed due to a positive drug screen.
Groups:
- All Consented Subjects: Of the 22 consented subjects, 15 screen-failed because prolactin levels did not meet eligibility criteria, and 1 screen-failed due to a positive drug screen. Because of this unanticipated high screen-failure rate, the study was terminated. Not enough subjects were randomized (N=6), or completed (N=5), to merit statistical analysis between study arms. Therefore, only the baseline characteristics of all consented/screened subjects (N=22) were published and are reported here.
Period: Overall Study
Arm/Group | All Consented Subjects
Started | 22
Completed | 5
Not Completed | 17
Not completed — Screen Fail | 16
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- All Consented Subjects: Of the 22 consented subjects, 15 screen-failed because prolactin levels did not meet eligibility criteria and 1 screen-failed due to a positive drug screen. Because of this unanticipated high screen-failure rate, the study was terminated. Not enough subjects were randomized or completed to merit statistical analysis between study arms. Therefore, only the baseline characteristics of all 22 consented/screened subjects were published and are reported here.
Arm/Group | All Consented Subjects
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.14 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Prolactin Levels for Individuals Treated With Adjunctive Amantadine Versus Placebo.
Time Frame: week 4 and week 8
Population: Of the 22 consented subjects, 15 screen-failed because prolactin levels did not meet eligibility criteria and 1 screen-failed due to a positive drug screen. Because of this unanticipated high screen-failure rate, the study was terminated. Only baseline characteristics of all 22 consented/screened subjects were published and are reported here.
Arm/Group | All Consented Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: entire study
Arm/Group | All Consented Subjects
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Too few subjects met study's eligibility criteria to run statistical analyses on primary outcomes. The baseline demographic data are reported here. Future research is needed to understand the prevalence of elevated prolactin in schizophrenia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes